CLINICAL TRIAL: NCT02835287
Title: Diabetes Complication Control in Community Clinics (D4C) Trial
Acronym: D4C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tulane University (Other)
Collaborators: Xiamen University (Other)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Chair, Tulane University Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 889920-1
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Hypertension; Dyslipidemia; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol-based Integrated Care (Experimental): The protocol-based integrated care, which will provide a standardized, combined, multi-component intervention according to clinical guideline treatment algorithms for diabetes and comorbidities in community clinics, will be delivered by care team (trained primary care physicians, health managers, and nurses supported by diabetes specialists) and assisted by a clinical decision support systems.
  Interventions: Other: Protocol-based integrated care
- Enhanced Control (Active Comparator): A usual team-based care delivered by trained primary care physicians, health managers, and nurses supported by diabetes specialists.
  Interventions: Other: Protocol-based integrated care

INTERVENTIONS:
Other: Protocol-based integrated care — The protocol-based integrated care, which will provide a standardized, combined, multi-component intervention according to clinical guideline treatment algorithms for diabetes and comorbidities in community clinics, will be delivered by trained primary care physicians, health managers, and nurses supported by diabetes specialists.

SUMMARY:
The overall objective of the proposed cluster randomized trial is to test whether implementation of protocol-based integrated care will improve CVD risk factors (glycated hemoglobin [HbA1C], systolic blood pressure [SBP], and LDL-cholesterol) over 18 months and reduce major CVD events (non-fatal stroke, non-fatal myocardial infarction, hospitalized heart failure, and CVD mortality) over 3 years among patients with type 2 diabetes and additional CVD risk factors or clinical CVD compared to usual team-based care in community clinics in Xiamen, China.

DETAILED DESCRIPTION:
Diabetes has reached epidemic proportions in China. Most patients with diabetes have multiple uncontrolled cardiovascular disease (CVD) risk factors due to suboptimal care, especially in underserved populations. The overall objective of the proposed cluster randomized trial is to test whether implementation of protocol-based integrated care (team-based care with clinical decision support systems) will improve CVD risk factors (glycated hemoglobin [HbA1C], systolic blood pressure [SBP], and LDL-cholesterol) over 18 months and reduce major CVD events (non-fatal stroke, non-fatal myocardial infarction, hospitalized heart failure, and CVD mortality) over 3 years among patients with type 2 diabetes and additional CVD risk factors or clinical CVD compared to usual team-based care in community clinics in Xiamen, China. The protocol-based integrated care, which will provide a standardized, combined, multi-component intervention according to clinical guideline treatment algorithms for diabetes and comorbidities in community clinics, will be delivered by trained primary care physicians, health managers, and nurses supported by diabetes specialists. The proposed trial will recruit approximately 12,160 patients with diabetes and additional CVD risk factors or clinical CVD from 38 community-based primary care clinics (community health service centers) in Xiamen, China. Nineteen community clinics with approximately 320 participants each will be randomly assigned to the intervention group and 19 community clinics with similar participants to the control group matched by administrative district and socioeconomic status. The protocol-based integrated care intervention will last for 36 months. HbA1C, BP, LDL-cholesterol, other variables, and co-morbidities will be measured at baseline and follow-up visits at months 6, 12, 18, 24, 30 and 36. In phase 1 (during the first 18-month intervention), the primary outcome is reduction in HbA1c, BP, and LDL-cholesterol measured by differences in mean changes in HbA1c, LDL cholesterol, and systolic BP levels over 18 months simultaneously modeled for a single overall treatment effect and proportion of patients with controlled HbA1c, BP, and LDL-C at 18 months. In phase 2 (during the three-year intervention), the primary outcome is the difference in major CVD incidence (non-fatal stroke, non-fatal myocardial infarction, hospitalized heart failure, and CVD mortality) between intervention and control groups. The secondary outcomes include: (1) the net changes in HbA1C, SBP, and LDL-cholesterol; (2) estimated 10-year risk of CVD; (3) the proportion of participants with controlled HbA1C, systolic BP, and LDL-cholesterol; (4) health-related quality of life; and (5) cost-effectiveness of intervention over three years. The proposed trial is designed to provide 90% statistical power to detect a 5% increase in the combined control rate of HbA1C, SBP, and LDL-cholesterol levels in phase 1 and a 20% reduction in major CVD (non-fatal stroke, non-fatal myocardial infarction, hospitalized heart failure, and CVD mortality) in phase 2 at a significance level of 0.05 for a two-sided test. This will be the first randomized cluster trial to test the implementation of a protocol-based integrated care program on multiple CVD risk factors and CVD events in diabetes patients who receive care from community clinics in China. This implementation research project has a high impact in public health because it will generate urgently needed data on an effective, practical, and sustainable intervention program aimed at reducing the CVD burden among diabetes patients in middle- and low-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥50 years who received primary care from the participating community clinics
* Uncontrolled diabetes (HbA1C ≥7% or ≥7.5% if with clinical CVD) with at least one additional CVD risk factor (SBP ≥140 and/or DBP ≥90 mm Hg and/or LDL-cholesterol ≥100 mg/dL) or clinical ASCVD (acute coronary syndromes, ischemic stroke, transient ischemic attack, or peripheral artery disease)

Exclusion Criteria:

* Patients with NYHA class II-IV heart failure, or receiving hemodialysis, or with contraindications to metformin or statin treatments
* Women who are pregnant or plan to become pregnant
* Patients who cannot be followed for 36 months (due to a health situation or migration)
* Patients who are unwilling or unable to give informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11132 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C, SBP, and LDL between intervention and control groups, simultaneously modeled using a scaled marginal model which allows estimation of a single overall treatment effect and combined control rate of HbA1c, SBP, and LDL | 18 months
  For patients younger than 65 years, HbA1c ≤7.0% or ≤8.0% in those with complications; for patients 65 years or older, HbA1c ≤7.5% or HbA1c ≤8.5% in those with complications; LDL-cholesterol <100 mg/dL; and blood pressure <140/90 mm Hg
Incidence of composite major cardiovascular disease events | Three years
  Non-fatal stroke, non-fatal myocardial infarction, hospitalized heart failure, and CVD mortality

SECONDARY OUTCOMES:
HbA1C | 18 months
  Net change in HbA1c or proportion of controlled HbA1c
SBP | 18 months
  Net change in SBP or proportion of controlled BP
LDL-cholesterol | 18 months
  Net change in LDL or controlled LDL
CVD risk score | 18 months
  10-year risk of CVD using ACC/AHA Risk Scores
Health-related quality of life: 12-item Short-Form Health Survey | Three years
  Health-related quality of life by the 12-item Short-Form Health Survey
Cost-effectiveness | Three years
  Incremental Cost-Effectiveness Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Study Chair — Tulane University
Locations (2):
- Tulane University, New Orleans, Louisiana, United States
- Xiamen Diabetes Institute, Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi X, He J, Lin M, Liu C, Yan B, Song H, Wang C, Xiao F, Huang P, Wang L, Li Z, Huang Y, Zhang M, Chen CS, Obst K, Shi L, Li W, Yang S, Yao G, Li X. Comparative Effectiveness of Team-Based Care With and Without a Clinical Decision Support System for Diabetes Management : A Cluster Randomized Trial. Ann Intern Med. 2023 Jan;176(1):49-58. doi: 10.7326/M22-1950. Epub 2022 Dec 6. PMID 36469915